CLINICAL TRIAL: NCT05756088
Title: The DEPICT Prospective Study: Determining the Association of Microvascular Disease as Assessed by PET and Graft Injury as Assessed by Donor Derived Cell Free DNA Post Transplantation
Brief Title: Determining the Association of Microvascular Disease as Assessed by PET and Graft Injury by Donor Derived Cell Free DNA
Acronym: DEPICT
Status: Withdrawn | Type: Observational
Why Stopped: Protocol was not approved by the sponsor; therefore PI not moving forward with this study.
Sponsor: Yale University (Other)
Collaborators: Yale Cardiovascular Research Group (Other); Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2000034497; YSI-004 (Other: Yale Cardiovascular Research Group)
Record Dates: First submitted 2023-02-22; First posted 2023-03-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Allograft Vasculopathy; Endothelial Dysfunction; Microvascular Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Low MFR (less than or equal to 1.5): Subjects who are found to have a low MFR of less than or equal to 1.5.
  Interventions: Diagnostic Test: Blood draw to measure the levels of dd-cf DNA
- Normal MFR (greater than 1.5): Subjects who are found to have normal MFR of greater than 1.5.
  Interventions: Diagnostic Test: Blood draw to measure the levels of dd-cf DNA

INTERVENTIONS:
Diagnostic Test: Blood draw to measure the levels of dd-cf DNA — Blood draw to measure the levels of dd-cf DNA.

SUMMARY:
The goal of this research study is to understand if a blood test in people who have had heart transplants can detect and predict the following:

* Blockages in the small blood vessels of the heart.
* Whether small blockages can turn into more severe blockages in the future.

Participants will undergo blood draws once every 3 months in the first year of the study (4 blood draws total, taking 15 minutes each) and their medical records will be reviewed for 3 years after the date they are enrolled in the study.

DETAILED DESCRIPTION:
A prospective, single center, assessment of donor derived cell free DNA in subjects who are post-heart transplant to assess correlation with microvascular flow as assessed by myocardial flow reserve (MFR) on positron emission tomography (PET).

Study design: This prospective, single center registry will enroll up to 88 subjects at Yale New Haven Health System (YNHHS). Patients who get PET scans for routine post-transplant surveillance will be included in the study. Up to an anticipated 44 subjects with low MFR and up to an anticipated 44 subjects with normal MFR will have dd-cf DNA drawn every 3 months for a year.

Patient population: A total of 88 adults referred to have an annual PET stress test as part of routine post-transplant surveillance for cardiac allograft vasculopathy and who are at least 3 years from heart transplantation and meet all eligibility criteria will be enrolled.

Diagnostic assessment: All subjects will have quarterly blood draws during the first year of enrollment to assess the levels of dd- cf DNA. All subjects will also undergo standard of care annual PET scans.

Subject follow up: All subjects will have routine follow-up as clinically necessary based on standard of care. Screening and follow-up data collection will occur through the electronic medical record.

Follow up duration: 3 years after enrollment.

Primary endpoint: Elevated dd-cf DNA levels in subjects with low MFR compared to normal MFR at up to one year follow-up post-enrollment.

Secondary Endpoints: The following secondary endpoints will be reported at 3 years post-enrollment based on the routine post-transplant standard of care:

* Combined clinical events of rejection, reduction in ejection fraction, need for revascularization, myocardial infarction, heart failure admissions and death or need for retransplantation.
* All-cause, cardiovascular, and non-cardiovascular mortality
* Myocardial infarction (Fourth Universal Definition)
* Revascularization (PCI or CABG)
* Hospitalization for heart failure
* Rejection
* Decrease in ejection fraction from baseline echo to 3 years follow up.
* Retransplantation

Procedure summary: Patients will undergo routine post-transplant surveillance and management per the discretion of the treating physician and per YNHHS post-heart transplant protocols. Quarterly study blood draws will be conducted in the first year of the study and will include dd-cf DNA measurements. These results will not be available to study team or the patients. All study participants will be blinded to these results.

ELIGIBILITY:
Potential subjects must meet all of the following criteria to be eligible for inclusion in the study:

General Inclusion Criteria:

* The patient is over 18 years of age.
* The patient underwent orthotopic heart transplantation and is undergoing routine cardiac allograft vasculopathy (CAV) surveillance with PET.
* The patient has no evidence of cardiogenic shock.
* The patient has no evidence of acute rejection.
* The patient, or legally authorized representative, has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent, approved by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC).

Potential subjects will be excluded if any of the following conditions apply:

Exclusion Criteria:

* Evidence of moderate to large area of ischemia on the PET.
* Multiorgan transplantation.
* Life expectancy <1 year due to non-cardiac conditions.
* Less than 3 years from transplantation.
* Patient appears unlikely or unable to participate in the required study procedures, as assessed by the study PI, study coordinator, or designee (ex: clinically-significant psychiatric, addictive, or neurological disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An anticipated total of 88 adults who are undergoing routine stress PET scans as part of post-transplant surveillance will be included. Patients who are at least 3 years from heart transplantation and who meet all eligibility criteria will be enrolled.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
dd-cf DNA and myocardial flow reserve (MFR) on positron emission tomography (PET) scan. | Baseline up to 1 year
  Changes in dd-cf DNA levels in subjects with low MFR compared to normal MFR.

SECONDARY OUTCOMES:
Impact of low MFR on rejection | 3 years
  Changes in rates of rejection in participants with low MFR compared with normal MFR.
Impact of low MFR on left ventricular ejection fraction | Baseline up to 3 years
  Changes in left ventricular ejection fraction in participants with low MFR compared with normal MFR.
Impact of low MFR on need for revascularization | 3 years
  Changes in rates of need for revascularization in participants with low MFR compared with normal MFR.
Impact of low MFR on myocardial infarction (MI) | 3 years
  Changes in rates of MI in participants with low MFR compared with normal MFR.
Impact of low MFR on admissions for heart failure | 3 years
  Changes in number of admissions for heart failure in participants with low MFR compared with normal MFR.
Impact of low MFR on retransplantation | 3 years
  Changes in rates of retransplantation in participants with low MFR compared with normal MFR.
Impact of low MFR on death | 3 years
  Changes in rate of death in participants with low MFR compared with normal MFR.

CONTACTS AND LOCATIONS:
Overall Officials: Lavanya Bellumkonda, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Health, New Haven, Connecticut, United States